CLINICAL TRIAL: NCT06444373
Title: Development of an Artificial Intelligence Model in Lung Cancer Screening for the Diagnosis of Lung Nodules and Risk Stratification in Subjects With Occupational and/or Smoking Exposure
Brief Title: Artificial Intelligence in Lung Cancer Screening
Acronym: INAIL BRIC
Status: Completed | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Giulia Veronesi, Medical Doctor, Scientific Institute San Raffaele
Other Study IDs: 116/INT/2022
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer Screening; Asbestos
Keywords: Artificial Intelligence; Asbestos; Lung Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects enrolled in lung cancer screening: Actual Smokers or formers smoker; Age > 50 years.

SUMMARY:
Single-center, non-profit, observational, retrospective study of collection of clinical and amnestic data and images to create, implement and develop a pilot model of an integrated virtual platform.

DETAILED DESCRIPTION:
The project we propose is a study whose objective was to develop an artificial intelligence program integrated into a web-based platform for the optimization of the performance of lung cancer screening for the diagnosis of lung nodules and risk stratification in subjects exposed to environmental carcinogens and/or cigarette smoke.

Inclusion criteria:

Age > 50; smokers for at least 20 pack-years (20 cigarillos a day for 20 years) or former heavy smokers if they quit less than 15 years ago; and/or previous professional exposure to asbestos; absence of lung cancer symptoms; who performed lung cancer screening after the year 2000 upon approval of the study by the relevant EC.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years;
* smokers for at least 20 pack-years (20 cigarettes a day for 20 years) or former heavy smokers if they quit less than 15 years ago;
* and/or previous professional exposure to asbestos;
* absence of lung cancer symptoms;
* who performed lung cancer screening after the year 2000 upon approval of the study by the relevant Etical Committee

Exclusion Criteria:

* Age < 50 years
* never smokers
* lung cancer symptoms

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age > 50 years; smokers for at least 20 pack-years (20 cigarettes a day for 20 years) or former heavy smokers if they quit less than 15 years ago; and/or previous professional exposure to asbestos.
  All subjects were enrolled in lung cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
AIM 1 Pilot deep learning model | from enrollment to the end of treatment at 2 years
  Development and fine-tuning of a pilot deep learning model for automatic detection and diagnosis of screen-detected nodules for risk stratification in subjects with asbestos exposure as part of a lung cancer screening program in high-risk subjects for exposure to asbestos and smoking on retrospective data.

SECONDARY OUTCOMES:
AIM 2 Clinical database | from enrollment to the end of treatment at 2 years
  Development of an integrated system between the clinical database and several existing imaging volumetric software and risk models for the creation of a pilot platform in order to optimize the organizational management of lung cancer screening.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy